CLINICAL TRIAL: NCT05893095
Title: Evaluation of Laparoscopic Peritoneal Lavage for Perforated Diverticulitis: A National Registry - Based Study
Status: Completed | Type: Observational
Sponsor: Uppsala University Hospital (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Christos Kollatos, MD, Uppsala University Hospital
Other Study IDs: 2021-01441
Record Dates: First submitted 2023-04-20; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Diverticular Disease of Colon; Diverticulitis, Colonic; Peritonitis; Gastrointestinal Diseases; Digestive System Disease
Keywords: Perforated diverticulitis; Purulent peritonitis; Laparoscopic peritoneal lavage
MeSH Terms: conditions — Diverticulosis, Colonic; Diverticulitis, Colonic; Peritonitis; Gastrointestinal Diseases; Digestive System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to study the emergency surgical treatment of diverticular disease in Sweden outside clinical trials. The main questions it aims to answer are:

* Which is the preferred surgical method of acute diverticular disease in Sweden?
* Which are the short and long-term outcomes of the different surgical methods?

Researchers will compare the different methods to see if there is a surgical operation that is superior for the treatment of acute diverticulitis.

DETAILED DESCRIPTION:
A retrospective study of patients who were admitted to a Swedish hospital between 1st July 2014 and 31st December 2020 with an ICD-10 code for diverticular disease of the large intestine (K57.2- K57.9) will be included. Patients who underwent procedures relevant to diverticulitis will be identified and therefore will be included. Procedures will be grouped into two categories: Laparoscopic peritoneal lavage (Group I), and sigmoid resection with or without stoma (Group II).

The cohort will be studied from 1st January 1997 until the index date aiming to assess comorbidities, previous abdominal surgeries, and admissions for diverticular disease. A Charlson Comorbidity Index (CCI) system adjusted for Swedish ICD-10 version will be used to calculate a composite score to reflect comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or older who were admitted to a Swedish hospital between 1st July 2014 and 31st December 2020 with an ICD-10 code for diverticular disease of the large intestine (K57.2- K57.9).
* Emergency admissions.
* Patients who underwent procedures relevant to diverticulitis.

Exclusion Criteria:

* Patients who were diagnosed with colorectal cancer before the index date.
* Patients with synchronous operations that are supposed to be irrelevant to acute diverticulitis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be based on a national cohort gathered from National Patient Register, the National Cancer Register and the Cause of Death Register, obtained by the Swedish National Board of Health and Welfare.
Sampling Method: Probability Sample
Enrollment: 52863 (Actual)
Dates: Start 2014-07-01; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Preferred operation for acute colonic diverticular disease | Up to 78 months
  Laparoscopic peritoneal lavage or sigmoid resection

SECONDARY OUTCOMES:
Crossover surgery | 1 day
  Crossover from laparoscopy to resection surgery
Reoperation | From date of inclusion until the date of the end of study or date of death from any cause, whichever came first, assessed up to 78 months
  Disease- associated reoperations involving the bowel or abdominal wall
Overall survival | From date of inclusion until the date of the end of study or date of death from any cause, whichever came first, assessed up to 78 months
Postoperative length of hospital stay | From date of inclusion until the date of discharge, assessed up to 78 months
Colorectal cancer diagnosis | From date of inclusion until the date of the end of study or date of death from any cause, whichever came first, assessed up to 78 months
Thirty-day postoperative mortality | Up 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Christos Kollatos, MD, Principal Investigator — Uppsala University Hospital, Sweden

IPD SHARING:
Plan to Share IPD: No